CLINICAL TRIAL: NCT05772065
Title: Evaluation of Clinical Practice Guidelines and Educational Decision-support Tools on Medical Trainees' Confidence With Latent Tuberculosis (LTBI) Testing and Treatment: A Randomized Trial
Brief Title: Clinical Practice Guidelines Versus Decision-support for Latent Tuberculosis Infection (LTBI) Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00376488
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Latent Tuberculosis
Keywords: Tuberculosis; Education
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDC/NTCA guidelines only (Active Comparator): The control group will have a link to US guidelines only and use it as a resource to answer the case vignettes.
  Interventions: Behavioral: CDC/NTCA guidelines only
- LTBI ASSIST and CDC/NTCA guidelines (Experimental): The intervention group will have a link to both US guidelines, and the LTBI-ASSIST tool as resources to answer the case vignettes.
  Interventions: Behavioral: LTBI ASSIST and CDC/NTCA guidelines only

INTERVENTIONS:
Behavioral: CDC/NTCA guidelines only — The control group will have a link to US guidelines only.
  Arms: CDC/NTCA guidelines only
Behavioral: LTBI ASSIST and CDC/NTCA guidelines only — The intervention group will have a link to both US guidelines, and the LTBI-ASSIST tool.
  Arms: LTBI ASSIST and CDC/NTCA guidelines

SUMMARY:
Latent Tuberculosis infection (LTBI) guidelines can be complex. LTBI-ASSIST is a web-based interactive tool to navigate US LTBI clinical practice guidelines in a patient-centered format that may guide clinical decision making around Latent TB care.

The research goal is to determine the difference in reported confidence among trainees that are not experts in LTBI care. The investigators further aim to assess if access to the LTBI-ASSIST tool improves clinical decision making in a series of simulated case scenarios containing guideline-derived, multiple choice items, as well as assess the efficiency in navigating the scenarios - measured by time to complete the survey.

The investigators proposed a randomized study design, in which an electronic survey/questionnaire with 4 case scenarios consisting of 14 multiple choice questions. Participants providing informed consent will be randomized to receiving access to either US Centers for Disease Control (CDC)/National Tuberculosis (TB) Controllers Association (NTCA) Guidelines or the LTBI-ASSIST online tool. Those in the experimental arm will further complete a 10 question System Usability Scale to assess usability of the LTBI-ASSIST tool.

All Johns Hopkins medical trainees and residents will be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Student at Johns Hopkins School of Medicine, or Medical trainee at Hopkins Hospital or Bayview Program

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Reported confidence with LTBI management [using a Likert scale questionnaire developed by study team] | 3 months
  The primary outcome will be the change in reported confidence with LTBI management, comparing between the control and intervention group. This outcome will be measured using a Likert Scale questionnaire administered pre- and post-intervention asking trainees to rate their confidence in performing critical LTBI care proficiencies.

SECONDARY OUTCOMES:
Proportion of appropriate LTBI care selection | 3 months
  The number of multiple choice questions answered correctly in the case scenarios comparing between trainees and/or CDC/NTCA guidelines.
Time to LTBI care selection | 3 months
  The time required for each group to reach a correct answer.

CONTACTS AND LOCATIONS:
Overall Officials: Maunank Shah, MD, PhD, Principal Investigator — Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Starke SJ, Martinez Rivera MB, Krishnan S, Shah M. Randomized Controlled Trial of Clinical Guidelines Versus Interactive Decision-Support for Improving Medical Trainees' Confidence with Latent Tuberculosis Care. J Gen Intern Med. 2024 May;39(6):951-959. doi: 10.1007/s11606-023-08551-3. Epub 2023 Dec 7. PMID 38062221